CLINICAL TRIAL: NCT07102849
Title: In-Depth Molecular Characterization in Marrow Failure Syndromes to Understand Clonal Dynamics and Expansion
Brief Title: Molecular and Clinical Analysis of Bone Marrow Failure: A Secondary Research Study
Status: Enrolling by invitation | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002422; 002422-H
Record Dates: First submitted 2025-08-02; First posted 2025-08-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-09-11

CONDITIONS: Bone Marrow Failure Disorders; VEXAS Syndrome; Hemoglobinurea, Paroxysmal; Myelodysplastic Syndromes; Bone Marrow Diseases
Keywords: Bone Marrow Failure; Aplastic Anemia; Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Bone Marrow Failure Disorders; VEXAS syndrome; Myelodysplastic Syndromes; Bone Marrow Diseases; Anemia, Aplastic; Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Biospecimens and data from age matched healthy volunteers (age 8 and up) will be used from the following protocol:- 07H0113 Procurement and Analysis of Blood, Bone Marrow, and Buccal Mucosa Samples from Healthy Volunteers to Support Clinical and Translational Research Projects in the NHLBI.
- Participants with Bone Marrow Failure Disorders: Biospecimens and data from children and adults with BMFS who participated in the following studies will be used:- 04H0012 "Collection of Tissue Specimens from Patients with Solid Tumors or Blood Disorders and Their HLA-Compatible Family Members"Clinical and research data from children and adults with BMFS who participated in the following studies will be used:- 06H0034 "Three Immunosuppressive Treatment Regimens for Severe Aplastic Anemia"- 12H0150 "Eltrombopag with Standard Immunosuppression for Severe Aplastic Anemia"- 20H0033 "Early Initiation of Oral Therapy with Cyclosporine and Eltrombopag for Treatment Naive Severe Aplastic Anemia (SAA)"- 09H0154 "A Pilot Study of the Thrombopoietin-Receptor Agonist Eltrombopag, in Refractory Aplastic Anemia Patients"

SUMMARY:
STUDY DESCRIPTION:

Bone marrow failure can result from immune mediated attack on stem cells or from inherited genetic defects such as telomere biology disorders or Fanconi anemia. Aplastic anemia (AA), a prototype of bone marrow failure syndromes (BMFS), can be acquired or inherited. Acquired BMFS have common immune mediated pathophysiology, and include AA, lower risk myelodysplastic syndrome (MDS, particularly hypoMDS), VEXAS, large granular lymphocytosis (LGL), paroxysmal nocturnal hemoglobinuria (PNH), pure red cell aplasia (PRCA), or cytopenia of undetermined origin. Clonality is frequent in patients with BMFS. Patients with acquired AA are known to have somatic mutations in phosphatidylinositol glycan class A (PIGA), BCL6 corepressor (BCOR) and HLA genes, which are all related to the immune mediated pathophysiology and good predictors of treatment and overall outcomes. Others such as ASXL1, RUNX1, and splicing factor mutations and/or chromosome 7 aneuploidy are associated with secondary myeloid neoplasms in these patients. Somatic mutations in STAT, DNMT3A and TET2 are prevalent in many other BMFS, such as LGL and VEXAS. Except for acquired AA, the clonal dynamics and trajectories, and cooccurrence of these aberrations in other BMFS are poorly understood. How these clonal events interact with epigenetic and proteomic changes are also unknown. In addition, the role of novel genetic defects in marrow failure is poorly characterized, such as mutations associated with inborn errors of immunity or complement pathways. Our aim is to elucidate this further using multi-omics, bulk/single cell DNA and RNA techniques as well as understand the epigenetics using ATAC-seq, and proteomics. The translation work will be correlated with clinical outcomes and laboratory parameters of patients with the particular BMFS cohort being investigated.

OBJECTIVES:

Primary Objective: To characterize the molecular aberrations in BMFS and to understand how clonality, epigenetics, and proteomics contribute to hematopoiesis over the course of disease using high resolution multi-omics characterization of hematopoietic stem and progenitor cells (HSPC), immune cells and other cellular composition in peripheral blood and bone marrow samples.

Secondary Objectives:

* To correlate the molecular findings with disease presentation and clinical outcomes (response to treatment, clonal evolution to secondary myeloid neoplasm, survival)
* To correlate molecular findings with clinical laboratory data, cytokine, chemokine, soluble receptor levels and growth factors
* To correlate findings with peripheral or marrow flow cytometry phenotyping
* To correlate findings on this study with already performed germline or somatic mutational data
* To compare the genomic, epigenomic and proteomic findings with healthy age matched controls

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

Bone marrow failure can result from immune mediated attack on stem cells or from inherited genetic defects such as telomere biology disorders or Fanconi anemia. Aplastic anemia (AA), a prototype of bone marrow failure syndromes (BMFS), can be acquired or inherited. Acquired BMFS have common immune mediated pathophysiology, and include AA, lower risk myelodysplastic syndrome (MDS, particularly hypoMDS), VEXAS, large granular lymphocytosis (LGL), paroxysmal nocturnal hemoglobinuria (PNH), pure red cell aplasia (PRCA), or cytopenia of undetermined origin. Clonality is frequent in patients with BMFS. Patients with acquired AA are known to have somatic mutations in phosphatidylinositol glycan class A (PIGA), BCL6 corepressor (BCOR) and HLA genes, which are all related to the immune mediated pathophysiology and good predictors of treatment and overall outcomes. Others such as ASXL1, RUNX1, and splicing factor mutations and/or chromosome 7 aneuploidy are associated with secondary myeloid neoplasms in these patients. Somatic mutations in STAT, DNMT3A and TET2 are prevalent in many other BMFS, such as LGL and VEXAS. Except for acquired AA, the clonal dynamics and trajectories, and cooccurrence of these aberrations in other BMFS are poorly understood. How these clonal events interact with epigenetic and proteomic changes are also unknown. In addition, the role of novel genetic defects in marrow failure is poorly characterized, such as mutations associated with inborn errors of immunity or complement pathways. Our aim is to elucidate this further using multi-omics, bulk/single cell DNA and RNA techniques as well as understand the epigenetics using ATAC-seq, and proteomics. The translation work will be correlated with clinical outcomes and laboratory parameters of patients with the particular BMFS cohort being investigated.

OBJECTIVES:

Primary Objective: To characterize the molecular aberrations in BMFS and to understand how clonality, epigenetics, and proteomics contribute to hematopoiesis over the course of disease using high resolution multi-omics characterization of hematopoietic stem and progenitor cells (HSPC), immune cells and other cellular composition in peripheral blood and bone marrow samples.

Secondary Objectives:

* To correlate the molecular findings with disease presentation and clinical outcomes (response to treatment, clonal evolution to secondary myeloid neoplasm, survival)
* To correlate molecular findings with clinical laboratory data, cytokine, chemokine, soluble receptor levels and growth factors
* To correlate findings with peripheral or marrow flow cytometry phenotyping
* To correlate findings on this study with already performed germline or somatic mutational data
* To compare the genomic, epigenomic and proteomic findings with healthy age matched controls

ELIGIBILITY:
* This study will utilize biospecimens and data with identifiers from up to 1,400 research participants with BMFS, aged 2 years and older, alongside age matched healthy volunteers aged 8 years and older.

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will utilize biospecimens and data with identifiers from up to 1,400 research participants with BMFS, aged 2 years and older, alongside age matched healthy volunteers aged 8 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2030-07-11 (Estimated); Study Completion 2030-07-11 (Estimated)

PRIMARY OUTCOMES:
Detection of molecular aberrations in marrow failure | baseline
  To characterize the molecular aberrations in marrow failure and to understand how clonality, epigenetics, and proteomics contribute to hematopoiesis over the course of disease using high resolution multi-omics characterization of HSPC, immune cells and other cellular composition in peripheral blood and bone marrow samples.

CONTACTS AND LOCATIONS:
Overall Officials: Bhavisha A Patel, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002422-H.html